CLINICAL TRIAL: NCT06814613
Title: The Effect of Progressive Relaxation Exercises Administered Via Telenursing on the Sleep Quality of Nursing Students After the Earthquake in Turkey
Brief Title: The Effect of Progressive Relaxation Exercises on the Sleep Quality of Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, seher ÇEVİK, Principal Investigator, Inonu University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: seher CEVİK AKTURA
Record Dates: First submitted 2025-01-25; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: University Students
Keywords: Earthquake; Nursing students; Progressive relaxation exercises; Sleep; Telenursing
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental model
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Progressive relaxation exercises were conducted by the researcher, who had received training in this area. The students were informed in detail about the study's implementation process.
  For the next 4 weeks, every night, 1 hour before the routine bedtime (or the time when the student planned to sleep), a video call (via the Google Meet application) was made with the student, and progressive relaxation exercises were performed. The exercise took approximately 20 minutes and followed the implementation protocol (Davis et al., 2008; Payne, 2000). Group interviews were conducted for students with similar sleep hours. They were asked to move to a ventilated room away from noise so that the exercises could be practiced comfortably and not interrupted.
  Interventions: Other: Exercise
- control (No Intervention): No intervention was applied to the control group in the study. Data collection forms were filled out only at the beginning and in the fourth week of the study.

INTERVENTIONS:
Other: Exercise — For the next 4 weeks, every night, 1 hour before the routine bedtime (or the time when the student planned to sleep), a video call (via the Google Meet application) was made with the student, and progressive relaxation exercises were performed. The exercise took approximately 20 minutes and followed the implementation protocol (Davis et al., 2008; Payne, 2000). Group interviews were conducted for students with similar sleep hours. They were asked to move to a ventilated room away from noise so that the exercises could be practiced comfortably and not interrupted.
  Other Names: Progressive relaxation exercises practice
  Arms: Intervention

SUMMARY:
Aim: The study aims to examine the effect of progressive relaxation exercises administered to nursing students via telenursing on sleep quality after the February 6 earthquake in Turkey.

Materials and Methods: The study was conducted as a randomized controlled study. The study population consisted of first-, second-, and third-year nursing students enrolled in the nursing departments of two universities located in eastern Turkey, who were residing in one of the 11 cities affected by the earthquake during the February 6 Turkey earthquake. The sample included 86 students (40 experimental, 46 control). While the control group received no intervention, the experimental group received progressive relaxation exercises for 20 minutes every night for 4 weeks, 1 hour before the routine bedtime (or the time they planned to go to sleep) by making a video call (via Google Meet application) with the student. Data were collected using a personal information form and the Pittsburgh Sleep Quality Scale. Descriptive statistical methods (frequency, percentage, arithmetic mean, standard deviation), independent groups t-test, and paired t-test were used to evaluate the data.

Conclusion: The research results can showed that progressive relaxation exercises could be an effective intervention in improving sleep quality after an earthquake. Additionally, conducting these exercises via telenursing could contribute significantly to the sustainability and control of the intervention.

DETAILED DESCRIPTION:
* If the students have any pre-sleep habits (using aromatic oil, massage, listening to music, etc.) that they routinely practice and that may affect the results of the study, they will be asked not to do so for 6 weeks.
* A video call is made with the students.
* The procedure is explained to the patient and any questions are answered or concerns are addressed.
* If possible, the patient is asked to move to a ventilated room away from noise so that the procedure can be performed comfortably and not interrupted.
* Procedure
* It is explained to the individual that the procedure can be done sitting or lying down and he/she is asked to release his/her muscles and take a comfortable position.
* The individual is asked to close his/her eyes and focus only on his/her body.
* For 5 seconds, the individual is asked to take a slow deep breath.
* He/she is asked to breathe out in a controlled manner in 3-4 seconds.
* The process of taking a deep breath in 5 seconds and giving it back in 3-4 seconds is repeated 3 times.
* While breathing, the individual is asked to squeeze his/her forehead muscles by raising his/her eyebrows as high as possible at the same time.
* After 10 seconds of tightening the forehead muscles, the patient is asked to slowly lower his/her eyebrows and slowly relax and release the forehead muscles while exhaling. He/she is encouraged to feel the relaxation in the forehead muscles.
* The individual is asked to take a deep breath, close his/her eyes tightly and squeeze the muscles around the eyes.
* After 10 seconds of tightening the muscles around the eyes, he/she is asked to slowly relax and release the muscles around the eyes while exhaling. With muscle

ELIGIBILITY:
Inclusion Criteria:

* The study included students who were in one of the 11 cities affected by the Turkey earthquake,
* did not have a medical diagnosis related to sleep disorders,
* were not using any sleep medications or long-acting treatments,
* had access to necessary equipment for telenursing such as the internet, computer, or phone,
* were enrolled in the first, second, or third year of the nursing program.

Exclusion Criteria:

* The fourth-grade nursing students were excluded from the study because they undergo internship training and work night shifts,
* which may affect their sleep patterns and quality and create a difference between them and other students.
* Students with any diagnosis related to sleep and those with any psychiatric diagnosis were also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | 3 month
  Pittsburgh Sleep Quality Index The scale was developed by Buysse et al. and validated in Turkish by Agargün et al. (Buysse et al., 1989; Agargün, 1996). Of the 24 items on the scale, 18 are included in the evaluation. The scale consists of 7 sub-dimensions: Subjective Sleep Quality, Sleep Latency, Sleep Duration, Habitual Sleep Efficacy, Sleep Disturbances, Use of Sleep Medication, and Daytime Dysfunction. Each sub-dimension is scored between 0-3, and the total scale score ranges from 0 to 21. An increase in the scale score indicates a decline in sleep quality. The results are evaluated in three categories: 0-5 points indicate healthy sleep, 6-10 points indicate poor sleep, and above 10 points indicate chronic sleep disturbance. The Cronbach's alpha internal consistency coefficient for the scale was calculated as 0.80 by Ağargün (1996).

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu university, Malatya, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Participants' data were collected for research purposes only according to the ethical principle of condentiality and protection. Therefore, it cannot be shared.